CLINICAL TRIAL: NCT05616676
Title: A Randomised Controlled Trial of a Brief Cognitive Task Intervention to Support NHS Staff Experiencing Intrusive Memories of Traumatic Events From Working in the COVID- 19 Pandemic.
Brief Title: A Brief Cognitive Task Intervention for NHS Staff Affected by COVID-19 Trauma (GAINS-2 Study)
Acronym: GAINS-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: P1vital Products Limited (Industry)
Collaborators: Wellcome Trust (Other); Uppsala University (Department of Psychology) (Unknown); Intensive Care Society (Communication Department) (Unknown); University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P1V-GAINS-IN02
Record Dates: First submitted 2022-11-11; First posted 2022-11-15 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Intrusive Memories of Traumatic Event(s)
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brief digital imagery-competing task (Experimental): Access to a brief digital imagery-competing task for 24 weeks (first 4 weeks with optional researcher support).
  Interventions: Behavioral: Brief digital imagery-competing task
- Brief digital music-listening task (Experimental): Access to a brief digital music-listening task for 24 weeks (first 4 weeks with optional researcher support).
  Interventions: Behavioral: Brief digital music-listening task
- Treatment As Usual (Experimental): Access to routine care that participants would otherwise receive if having intrusive memories of traumatic events for 24 weeks.
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Behavioral: Brief digital imagery-competing task — First session guided by a researcher: A memory cue followed by playing a computer game with mental rotation instructions.
  Option to engage in self-administered/guided sessions after the first session.
  Arms: Brief digital imagery-competing task
Behavioral: Brief digital music-listening task — First session guided by a researcher: Information about the composer's music followed by listening to classical music.
  Option to engage in self-administered/guided sessions after the first session.
  Arms: Brief digital music-listening task
Other: Treatment As Usual — Access to routine care that participants would otherwise receive if having intrusive memories of traumatic events.
  Arms: Treatment As Usual

SUMMARY:
Frontline healthcare staff are frequently exposed to traumatic events at work (e.g., witnessing patients die), amplified by the COVID-19 pandemic. A significant proportion experience intrusive memories of these events that pop suddenly into mind: they can disrupt functioning and can contribute to post-traumatic stress disorder. Previous research has shown that a brief behavioural intervention can reduce the number of intrusive memories after a traumatic event. In this study we will test the effect of a digital imagery-competing task, a digital music-listening task and treatment as usual (TAU) for National Health Service (NHS) staff with intrusive memories of work-related traumatic events from the pandemic. We test the effect on the number of intrusive memories (primary outcome), and other clinical symptoms (PTSD, anxiety, depression, and insomnia), in addition to work functioning, general functioning and quality of life (secondary outcomes). Intervention feasibility, acceptability and implementation will also be explored (additional outcomes). We will recruit approximately 150 NHS staff (via the Intensive Care Society, social media and direct advertising by NHS Trusts) with intrusive memories of traumatic events experienced during the COVID-19 pandemic.

The study is funded by the Wellcome Trust (223016/Z/21/Z).

DETAILED DESCRIPTION:
A statistical analysis plan will be prepared prior to the first interim analysis using Bayesian analyses for statistical inference.

Regular monitoring will be performed by P1vital Products to verify that the study is conducted, and data are generated, documented and reported in compliance with the protocol, GCP and the applicable regulatory requirements. Quality assurance representatives from the Sponsor may carry out an audit of the study in compliance with regulatory guidelines and relevant standard operating procedures.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above.
* Able to read, write and speak in English.
* Worked in a clinical role with COVID-19 patients in the NHS during the COVID-19 pandemic.
* Experienced at least one traumatic event related to their clinical work during the COVID- 9 pandemic meeting criterion A of the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria for Post-Traumatic Stress Disorder (PTSD): "exposure to actual or threatened death, serious injury, or sexual violence" by "directly experiencing the traumatic event(s)" or "witnessing, in person, the event(s) as it occurred to others".
* Experience intrusive memories of the traumatic event(s).
* Experienced at least three intrusive memories in the week prior to screening.
* Have internet access.
* Willing and able to provide informed consent and complete study procedures
* Willing and able to be contacted by the research team during the study period.
* Have not taken part in a previous study of this intervention from this research team

Exclusion Criteria:

• Have fewer than three intrusive memories during the run-in week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Number of intrusive memories of traumatic event(s) | Week 4 (all arms) controlling for run-in/baseline week
  Number of intrusive memories of traumatic event(s) recorded by participants in a brief daily online diary for 7 days.

SECONDARY OUTCOMES:
Number of intrusive memories of traumatic event(s) | Weeks 12 and 24 (all arms) controlling for run-in/baseline week
  Number of intrusive memories of traumatic event(s) recorded by participants in a brief daily online diary for 7 days.
PTSD Checklist for DSM-5 (PCL-5) | Baseline, 4 weeks, 12 weeks and 24 weeks (all arms)
  This 20-item measure assesses symptoms of PTSD over the last week. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Scores are summed to give a total severity score (ranging 0 to 80).
Sleep Condition Indicator (SCI) | Baseline, 4 weeks, 12 weeks and 24 weeks (all arms)
  This 2-item scale measures sleep problems against the DSM-5 criteria for insomnia disorder. Item responses are each scored 0-4, with scores from 0 to 2 indicating threshold criteria for insomnia disorder. Total score ranges 0-8, with a higher score indicating better sleep.
Generalised Anxiety Disorder 2-item scale (GAD-2) | Baseline, 4 weeks, 12 weeks and 24 weeks (all arms)
  This 2-item short-form self-report measure assesses symptoms of anxiety. Items are rated for how often they have bothered the respondent over the last two weeks, from 0 ("not at all") to 3 ("nearly every day"). Total score is the sum of both items and ranges from 0 to 6.
Patient Health Questionnaire 2-item version (PHQ-2) | Baseline, 4 weeks, 12 weeks and 24 weeks (all arms)
  This 2-item short-form self-report measure assesses symptoms of depression. Items are rated for how often they have bothered the respondent over the last two weeks, from 0 ("not at all") to 3 ("nearly every day"). Total score is the sum of both items and ranges from 0 to 6.
Scale of Work Engagement and Burnout (SWEBO) | Baseline, 4 weeks, 12 weeks and 24 weeks (all arms)
  This 19-item self-report measure assesses work engagement and burnout. The work engagement subscale consists of 10 items assessing three dimensions (vigour, attentiveness, dedication). The burnout subscale consists of 9 items assessing three dimensions (exhaustion, disengagement and inattentiveness). Respondents rate how often they have felt each descriptive in the past two weeks, from 1 (not at all) to 4 (all the time). The mean score is calculated for each subscale.
Sickness absence | Baseline, 4 weeks, 12 weeks and 24 weeks (all arms)
  Single item assessing self-reported number of sick days taken from work in the last 4 weeks.
Intention to leave job | Baseline, 4 weeks, 12 weeks and 24 weeks (all arms)
  3 items assess participants' intention to leave their job e.g. "I think a lot about leaving the job", each rated from 1 (strongly agree) to 5 (strongly disagree). The total score ranges 3 to 15, with a lower score indicating stronger intention to leave the job.
5-level European Quality of Life 5 Dimension (EQ-5D-5L) | Baseline, 4 weeks, 12 weeks and 24 weeks (all arms)
  The 5-level version of the EuroQol-5D (EQ-5D-5L) is a brief measure for assessing general quality of life and health status. Items assess mobility, self-care, usual activities, pain/discomfort and anxiety/depression each on a 5-point scale. 5 items are scored on a 5-point ordinal scale from 'no problem' (1) to 'highest level of problems' (5). Respondents also rate their overall health today from 0 (the worst health you can imagine) to 100 (the best health you can imagine). Scores are analysed separately (not summed).
World Health Organization Disability Assessment Schedule 12-item version (WHODAS 2.0) | Baseline, 4 weeks, 12 weeks and 24 weeks (all arms)
  The 12-item, self-report version of the WHODAS 2.0 will be used to assess difficulties in relation to the impact of intrusive memories. Respondents rate how much difficulty they have had in each area in the past 30 days, from 0 (none) to 4 (extreme or cannot do). The overall score is calculated as a percentage of the maximum possible score (i.e., 48 points).
Intrusive memory ratings | Baseline, 4 weeks, 12 weeks and 24 weeks (all arms)
  The 9-item questionnaire assesses a number of intrusive memories characteristics. These characteristics include frequency (7-point categorical response from 'never' to 'many times a day'); distress (0=not at all to 10=extremely); disruption to concentration (0=not at all to 10=extremely); interference with what you were doing (how much (0=not at all to 10=extremely) and for how long (6-point categorical response from '<1min' to '>60mins')); impact on work functioning (how much (0=not at all to 10=extremely) and in what ways (open text response)); impact on functioning in other areas of life (how much (0=not at all to 10=extremely) and in what ways (open text response)).

OTHER OUTCOMES:
Changes to health and work | 4 weeks, 12 weeks and 24 weeks (all arms)
  The 9-item questionnaire will be used to assess the occurrence and number of any new traumatic events, any additional stressful life events (e.g. relationship problems, financial problems), new treatments received, untoward medical occurrences, changes to the job, or changes to the number of hours worked per week since the last assessment.
Feedback questionnaire | After 4 weeks (brief imagery-competing task and brief music listening task arms only)
  A 12-item questionnaire assessing participants' experience of using the brief cognitive task. The first ten items assess how easy, helpful, distressing, burdensome and acceptable participants found the brief cognitive task, how willing they would be to use it in the future, how confident they would be in recommending it to a friend and how much they feel it could be used to support staff within the NHS, each rated from 0 (not at all) to 10 (very). The last two items ask how the brief cognitive task could be improved, and for any other comments or suggestions about the brief cogntive task, both with an open response.
Optional qualitative interview | At 4 weeks and at 12-24 weeks (brief imagery competing task and brief music listening task arms only)
  This semi-structured interview will consist of a number of questions designed to gain an in-depth understanding of participants' experience of using the brief cognitive task, including acceptability, improvement suggestions, and potential barriers/facilitators to implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Holmes, Principal Investigator — Uppsala University (UU), Sweden
Locations (1):
- P1vital Products Ltd, Wallingford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The Study Protocol and Statistical Analysis Plan will be shared on the Open Science Framework, together with an anonymised database of individual participant data, data dictionary, and analysis scripts.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The Study Protocol and Statistical Analysis Plan were uploaded to the Open Science Framework (OSF) prior to the last participant completing the last visit.
  Results of the study will be shared through open access publications. On publication of the main study results, the associated database of individual participant data (anonymised), data dictionary, and analysis scripts will be made available on OSF.
  The information described above will be shared indefinitely and with no end date on the OSF platform.
Access Criteria: The information described above will be made available on the OSF indefinitely.
  OSF is an open source web application that is freely accessible to the public and scientific community.
URL: https://osf.io/cs6hn/